CLINICAL TRIAL: NCT04199832
Title: Nutritional Status and Complications in Patients Undergoing Chemoradiotherapy for Esophageal Squamous Cell Carcinomas: a Comparison of Nasogastric Tube, Percutaneous Endoscopic Gastrostomy Tube and Oral Supplement
Brief Title: To Compare the Effect of Different Nutritional Pathways on Improving Nutritional Status of Esophageal Cancer Patients Undergoing Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20190920
Record Dates: First submitted 2019-12-02; First posted 2019-12-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Enteral Nutrition
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nasogastric tube: The patient had difficulty swallowing before chemoradiotherapy and placed a nasogastric tube.
  Interventions: Dietary Supplement: Dietary guidance
- gastrostomy feeding: Patients with dysphagia before chemoradiotherapy began to voluntarily choose gastrostomy feeding.
  Interventions: Dietary Supplement: Dietary guidance
- Oral intake: Patients with normal swallowing or not receiving tube feeding.
  Interventions: Dietary Supplement: Dietary guidance

INTERVENTIONS:
Dietary Supplement: Dietary guidance — Dietary guidance for feeding tube patients with food homogenate，dietary guidance for patients with oral feeding.

SUMMARY:
This study prospectively recruited esophageal squamous-cell carcinoma patients who received nasogastric tube (NG), gastrostomy feeding and oral intake to compare the changes in nutritional status and quality of life during chemoradiation therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically proven esophageal squamous cell carcinoma
* Karnofsky performance score(KPS) ≧70
* Concurrent chemoradiotherapy
* Hemoglobin≥90.0g/dL,white blood cell count（WBC）≥ 4000 cells/mm³,Platelet count≥100,000 cells/mm³
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal,bilirubin normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Patients have good compliance to treatment and follow-up of acceptance
* the functions of the heart, kidney, liver were basically normal, with no chemotherapy and radiotherapy contraindications

Exclusion Criteria:

* Patients with severely bowel function impaired or can not tolerate enteral nutrition
* Patients with serious gastrointestinal obstruction, be unable to take food by mouth and can not / do not want to a feeding tube inserted
* Patients who have severe vomiting, gastrointestinal bleeding, intestinal obstruction
* Patients who have distant metastasis
* The primary tumor or lymph node already received surgical treatment efuse or incapable to sign the informed consent form of participating this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal squamous cell carcinoma who received concurrent chemoradiotherapy voluntarily chose different nutritional treatment paths according to the degree of dysphagia.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Body Weight Change from baseline to the end of treatment | up to 1 month after the treatment
  Body weight change from baseline to the end of treatment = body weight at the end of treatment - baseline body weight.

SECONDARY OUTCOMES:
Blood biochemical examination | up to 1 month after the treatment
  albumin,prealbumin,haemoglobin,et al, record the changes before and after the treatment.
Scored Patient-Generated Subjective Global Assessment (PG-SGA) | up to 1 month after the treatment
  Nutritional status evaluation table. score: 0-1 A: well-nourished; score：2-8 B: moderately malnourished; score：≥9 C: severely malnourished.
EORTC QLQ-C30 | up to 1 month after the treatment
  Quality of life evaluation form. QLQ-C30 results were linearly transformed to scores 0 to 100. Higher scores represent worse symptoms in the symptom scales and better function in functional scales.
Grade 3-5 toxicity | up to 1 month after the treatment
  Grade 3-5 adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 andthe criteria of the Radiation Therapy Oncology Group ，such as esophagitis、pneumonitis 、hematologic toxicity and infection rate
Completion rate of chemoradiotherapy | up to 1 month after the treatment
  The proportion of people who complete all treatment as required
Overall Survival | at least 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Qingsong Pang, Doctor, Study Chair — Department of Radiation Oncology,Tianjin Medical University cancer Institute and Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Dong J, Dai Z, Cao F, Zhang W, Zhang T, Chen X, Chen Y, Zhao F, Li J, Du Q, Zhang K, Zeng Y, Li C, Wang Y, Li Y, Wang K, Pang Q. Effects of PEG in patients with esophageal squamous cell carcinoma during concurrent chemoradiotherapy: a prospective study. Gastrointest Endosc. 2023 Dec;98(6):901-910.e3. doi: 10.1016/j.gie.2023.04.2094. Epub 2023 May 5. PMID 37150411